CLINICAL TRIAL: NCT05278221
Title: Development and Optimization of Transcranial Magnetic Stimulation (TMS) Combined With EEG/EMG as a Biomarker Predicting Response to Antiepileptic Drugs
Brief Title: TMS Combined With EEG/EMG as a Biomarker Predicting Antiepileptic Drug Response
Acronym: BIOEPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BIOEPI
Record Dates: First submitted 2022-02-10; First posted 2022-03-14 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Focal Epilepsy
Keywords: epilepsy, medical device
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Intervention Model Description: The study has 2 parts; part I that includes healthy volunteers and part II that includes patients with focal epilepsy. Each healthy volunteer will participate in three sessions every 2 weeks and will receive a single per os dose of Lacosamide (200 mg), Brivaracetam (50 mg) or placebo. Patients in part II will receive either Lacosamide, 300 mg p.o. or Brivaracetam, 100 mg p.o. All participants will perform a test using the tested software that combines a Transcranial Magnetic Stimulation with EEG/EMG
Who Masked: Outcomes Assessor
Masking Description: The evaluator of the outcomes will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Other): Each healthy volunteer during Part I of the study will receive every 2 weeks a single per os dose of Lacosamide (200 mg), Brivaracetam (50 mg) or placebo. All healthy volunteers will perform tests using the new software that combines Transcranial Magnetic Stimulation Combined With EEG/EMG,
  Interventions: Device: Software EstimLT
- Patients with focal epilepsy (Other): Patients during Part II, will receive the treatment according to the treating physician's discretion, regardless of the protocol, either with Lacosamide, 300 mg p.o. or Brivaracetam, 100 mg p.o. All patients will perform tests using the new software that combines Transcranial Magnetic Stimulation Combined With EEG/EMG,
  Interventions: Device: Software EstimLT

INTERVENTIONS:
Device: Software EstimLT — Healthy volunteers will receive a single per os dose of Lacosamide (200 mg), Brivaracetam (50 mg) or placebo and then the software will be tested

SUMMARY:
Ιn the present study (BIOEPI), the following three hypotheses will be investigated:

1. The proposed TMS-EEG / EMG protocol (which includes software for calculating the cerebral cortex stimulation threshold) in combination with advanced signal analysis and data mining methods will allow the detection of the effect of antiepileptic drugs (AED) with different mechanisms of action (lacosamide & brivaracetam) in the Central Nervous System under healthy and pathological conditions (Epilepsy).
2. AED-induced changes in selected TMS-EEG / EMG features predict the clinical response of individual epileptic patients to AED.
3. AED-induced changes in selected TMS-EEG / EMG features may predict cognitive side effects.

DETAILED DESCRIPTION:
The overarching objective of this study is to develop a combined TMS-EEG/EMG protocol so as to explore the effects of AEDs on cortical excitability and obtain novel electrophysiological biomarkers which could help predict the response of epileptic patients to AEDs, in line with the principles of personalized medicine. In order to achieve the overarching objective, we will perform a Diagnostic Clinical Performance Study, (FDA 2013) with the following specific objectives.

Primary Objective 1: To investigate whether TMS-EEG/EMG biomarkers can predict the response of patients with focal epilepsy to AEDs (Lacosamide & Brivaracetam).

Secondary Objective 1: Development, testing and validation of novel TMS-EEG/EMG stimulation and multi-level data analysis protocols, incorporating advanced methods of signal analysis, connectivity, complexity, and propagation across the cortical mantle.

Secondary Objective 2: Investigating the sensitivity of TMS-EEG/EMG biomarkers for detecting changes in brain physiology in healthy subjects and patients with focal epilepsy.Secondary Objective 3: Investigating whether TMS-EEG / EMG biomarkers may predict cognitive deficits in patients with focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

1. Adult volunteers aged 18-65 years
2. Able to provide informed consent
3. Meet the criteria of the attached TMS safety questionnaire (Rossi et al, 2011). It is clarified that: a) criterion 1 does not apply to the group of patients and b) a positive answer to criteria 5, 6, 8, 9 & 10 excludes inclusion in the study while the other answers are evaluated by the investigator.

Specific criteria:

The specific criteria per group of study participants are as follows:

Patient Group:

1. Adult patients, 18-65 years of age, suffering from focal epilepsy, as evidenced by clinical and EEG features.
2. All patients continue suffering from seizures despite treatment with 1-2 concomitant AEDs (with vagal nerve stimulation counting as an AED). In order to be eligible, patients should be suffering from simple partial seizures (SPS) and a motor component or complex partial seizures (CPS) with or without secondary generalization (sGS). Patients should report at least three seizures during the 12 weeks of Historical Baseline.
3. Patients are required to be Lacosamide and Brivaracetam-naive and, in the latter case, not taking concomitant Levetiracetam.
4. Patients are about to commence treatment with Lacosamide or Brivaracetam, as per the treating physician's orders. It is stressed that the decision to prescribe Lacosamide or Brivaracetam is made by the patient's treating physician totally independently from participation in the current study.
5. Epilepsies of genetic or unknown aetiology (patients with hippocampal sclerosis can be included). The epileptic patients will be a convenience sample recruited at the Epilepsy Outpatient Clinic of the University General Hospital of Thessaloniki "AHEPA".

Healthy control group:

Adult, healthy volunteers, 18-65 years of age

Exclusion Criteria:

The specific criteria per group of study participants are as follows:

Patient Group:

1. The presence of Central Nervous System "CNS" disorders other than epilepsy on history or examination
2. Comorbid psychiatric or medical conditions that may compromise the ability of the individuals to participate in the study
3. EEG evidence of generalized epilepsy.
4. Uncountable seizures due to clustering.
5. Use of centrally acting drugs other than AEDs.
6. Pregnancy or planned pregnancy prior to the index test.

Healthy control group:

1. Presence of medical or psychiatric conditions that may interfere with the procedures.
2. Contraindications to TMS (i.e. pregnancy, presence of heart pacemakers, metal objects etc).
3. History of adverse reactions to pharmacological agents.
4. History of alcohol or nicotine abuse or use of any other centrally acting drug.
5. Participation in another clinical trial in the previous 8 weeks.
6. Pregnancy or planned pregnancy prior to the index test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of TMS Combined With EEG/EMG for predicting response to AEDs | 9 months
  The Primary Outcome Measure is the diagnostic accuracy (calculated as the number of true positives + true negatives)/(number of true positives + true negatives + false positives + false negatives) of the index test for predicting response to AEDs (defined as reduction of seizure frequency by 50% or more during the maintenance period in comparison to baseline).
  The primary efficacy endpoint will be assessed in the combined groups of responders (LAC+BRV) and non-responders (LAC+BRV) because the starting hypothesis is that response to AEDs will be associated with alterations in TMS-EEG/EMG biomarkers.

SECONDARY OUTCOMES:
PPV, NPV, LR+ & LR- of TMS Combined With EEG/EMG for predicting response to AEDs | Through study completion, an average of 2 years
  Positive Predictive Value (PPV), Negative Predictive Value (NPV), positive likelihood ratio (LR+) & negative likelihood ratio (LR-) of TMS Combined With EEG/EMG for predicting response to AEDs (defined as reduction of seizure frequency by 50% or more).
Accuracy, PPV, NPV, LR+ & LR- of TMS Combined With EEG/EMG for other measures of response to AEDs | Through study completion, an average of 2 years
  Accuracy, PPV, NPV, positive likelihood ratio (LR+) & negative likelihood ratio (LR-) of TMS Combined With EEG/EMG for other measures of response to AEDs (i.e. percent seizure reduction, seizure freedom, time to n th (n=1,5th,10th) seizure).
Accuracy of TMS Combined With EEG/EMG for predicting AED-induced side-effects | Through study completion, an average of 2 years
  Accuracy of TMS Combined With EEG/EMG for predicting AED-induced cognitive side-effects and other study-emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Vasilios Kimiskidis, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No